CLINICAL TRIAL: NCT04333862
Title: Assessment of Covid-19 Infection Rates in Healthcare Workers Using a Desynchronization Strategy
Acronym: Covid-19
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-00563
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: SARS-CoV-2
Keywords: SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of nasal swabs twice per week and blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthcare workers providing healthcare: To determine the infection rate of healthcare workers providing healthcare versus those who are staying at home, in a desynchronization work strategy
- Healthcare workers staying at home: To determine the infection rate of healthcare workers providing healthcare versus those who are staying at home, in a desynchronization work strategy
- Hospitalized patients: To compare the infection rate of hospitalized patients versus healthcare workers

SUMMARY:
Desynchronization of infection rates in healthcare workers will potentially reduce the early infection rates and therefore maintain workforce for late time points of the epidemic. Given the current threat of the COVID-19 epidemic, the department for Visceral Surgery and Medicine, Bern University Hospital, has decided to limit its elective interventions to oncological and life-saving procedures only. At the same time, the medical team were split in two teams, each working for 7 days, followed by 7 days off, called a desynchronization strategy. Contacts between the two teams are avoided.

The main aim of present study is to determine, if the infection rate between the two populations (at work versus at home) is different. Secondary aims are to determine if the workforce can be maintained for longer periods compared standard of care, and if the infection rate among patients hospitalized for other reasons varies compared to the community.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) spreads rapidly and causes a pandemic of coronavirus disease 2019 (COVID-19, the disease caused by SARS-CoV-2). Protecting and supporting caregivers is essential to maintain the workforce in the hospital to treat patients.

The use of recommended barrier precautions such as masks, gloves and gowns is of highest priority in the care of all patients with respiratory symptoms. However, given the long incubation period of 5 days there will be undiagnosed but infected patients with clinically mild cases, atypical presentations or even no symptoms at all. Thus, healthcare workers are on the one side at risk to get infected by asymptomatic patients and on the other side are critically needed for later phases of the epidemic, when the resources will in all likelihood be scarce or depleted.

One potential strategy to maintain workforce throughout an epidemic is to reduce the workforce in the early phases. Reducing workforce at early phases might potentially reduce in-hospital infection of the caregivers and reduces early burnout. One way of reducing the active workforce is to postpone all elective and non-urgent medical interventions to later phases of the epidemic.

Desynchronization of infection rates in healthcare workers will potentially reduce the early infection rates and therefore maintain workforce for late time points of the epidemic. Given the current threat of the COVID-19 epidemic, the department for Visceral Surgery and Medicine, Bern University Hospital, has decided to limit its elective interventions to oncological and life-saving procedures only. At the same time, the medical team were split in two teams, each working for 7 days followed by 7 days off, called a desynchronization strategy. Contacts between the two teams are avoided. This new regulation took effect on March 16th 2020.

Currently available resources to perform tests for SARS-CoV-2 infection are limited for the clinical routine and are therefore not available for research purposes. Thus, in the context of a clinical study the investigators aim to perform additional testing of SARS-CoV-2 of healthcare workers and patients in order to determine the clinical consequences of such desynchronization strategy, firstly within the current epidemic and secondly for future outbreaks.

The main aim of present study is to determine if the infection rate between the two populations (at work versus at home) is different. Secondary aims are to determine if the workforce can be maintained for longer periods compared standard of care, and if the infection rate among patients hospitalized for other reasons varies compared to the community.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers of the Department for Visceral Surgery and Medicine
* Patients of the Department for Visceral Surgery and Medicine
* Written informed consent

Exclusion Criteria:

* No informed consent
* Patients with known COVID-19 infection before hospitalization in the investigators' department

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health care workers and patients of the Department for Visceral Surgery and Medicine
Sampling Method: Non-Probability Sample
Enrollment: 519 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Fraction of healthcare workers infected with SARS-CoV-2 | 90 days
  To determine the infection rate of healthcare workers providing healthcare versus those who are staying at home, in a desynchronization work strategy

SECONDARY OUTCOMES:
Fraction of healthcare workers with COVID-19 | 90 days
  To compare the infection rate of hospitalized patients versus healthcare workers
Number of patients infected in the hospital | 90 days
  Tracing origins of infection in healthcare workers to distinguish between community versus hospital acquired.
Development of SARS-CoV2 specific antibody repertoire | 18 months
  To determine the T and B cell specific antibody repertoire in the course of a COVID-19 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, Prof. Dr., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- Guido Beldi, Bern, Switzerland